CLINICAL TRIAL: NCT02036658
Title: fMRI of Emotion Regulation During RCT of CBT vs. MBSR for Social Anxiety Disorder
Brief Title: Emotion Regulation During RCT of CBT vs. MBSR for Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, James J. Gross, Professor of Psychology, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CBT-MBSR 10521038; R01MH076074 (NIH)
Record Dates: First submitted 2014-01-10; First posted 2014-01-15 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Social Anxiety Disorder
Keywords: social anxiety; treatment; cognitive-behavioral therapy; mindfulness-based stress reduction; emotion regulation; randomized controlled trial; neuroimaging; functional magnetic resonance imaging; mediators; mechanisms
MeSH Terms: conditions — Phobia, Social; Emotional Regulation | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: To investigate treatment outcome and mediators of Cognitive-Behavioral Group Therapy (CBGT) vs. Mindfulness-Based Stress Reduction (MBSR) vs. Waitlist (WL) in patients with generalized social anxiety disorder (SAD), unmedicated patients with a primary diagnosis of Social Anxiety Disorder (SAD) will be randomized to CBGT vs. MBSR vs. WL and will complete assessments at baseline, post-treatment/WL, and at 1-year follow-up, including the Liebowitz Social Anxiety Scale - Self-Report (primary outcome; Liebowitz, 1987) as well as measures of treatment-related processes.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive Behavioral Group Therapy (Active Comparator): Cognitive behavioral group therapy (CBGT) will be delivered by two Ph.D. clinical psychologists trained by Dr. Richard Heimberg to implement his CBGT for SAD (Heimberg & Becker, 2002). Groups of six individuals will meet for 12 sessions of 2.5 hours each. The participants will also use selected portions of the client workbook developed by (Hope, Heimberg, & Turk, 2010) to supplement relevant portions of the protocol. The treatment will be comprised of four major components: (1) psychoeducation and orientation to CBGT; (2) cognitive restructuring skills; (3) graduated exposure to feared social situations, within session and as homework; and (4) relapse prevention and termination. Further details of the treatment are available elsewhere (Heimberg & Becker, 2002).
  Interventions: Behavioral: Cognitive Behavioral Group Therapy
- Mindfulness-Based Stress Reduction (Active Comparator): MBSR will follow the standard curriculum outline compiled in 1993 by Jon Kabat-Zinn except that the one-day meditation retreat will be converted to four additional weekly group sessions between the standard class 6 and 7 so that there will be 12 weekly 2.5 hour sessions. This will be done to match the CBGT protocol in duration and time. The MBSR intervention will be delivered by a University of Massachusetts Center for Mindfulness certified MBSR instructor with more than 30 years of teaching experience. To support the practice, each participant will be given A Mindfulness-Based Stress Reduction Workbook (Stahl & Goldstein, 2010), which includes descriptions of mindfulness exercises together with pre-recorded audio files to support ongoing practice.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Waitlist Control (No Intervention): This will be a delayed treatment arm. Participants randomized to the waitlist control group will be re-randomized after completing the no treatment period of 12 weeks to CBGT or MBSR with equal probability.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Group Therapy — Cognitive Behavioral Group Therapy for social anxiety disorder is a 12-week treatment that involves psychoeducation, cognitive restructuring and exposure to social situations.
  Other Names: CBGT
  Arms: Cognitive Behavioral Group Therapy
Behavioral: Mindfulness-Based Stress Reduction — Mindfulness-Based Stress Reduction will be completed in 12 weeks in the study and includes enhancing one's awareness non-judgmentally by focusing on the present moment through the use of mindfulness meditation.
  Other Names: MBSR
  Arms: Mindfulness-Based Stress Reduction

SUMMARY:
The purpose of the study is to investigate the immediate and longer-term impact of Cognitive-Behavioral Group Therapy (CBGT) versus Mindfulness-Based Stress Reduction (MBSR) for patients with Social Anxiety Disorder.

DETAILED DESCRIPTION:
A. Aims

The overall goal of this research is to elucidate the neural bases of two specific forms of emotion regulation - cognitive regulation (CR) and attention regulation (AR). CR and AR are thought to be important mechanisms underlying therapeutic change associated with Cognitive-Behavioral Therapy (CBT) and Mindfulness-Based Stress Reduction (MBSR) for generalized Social Anxiety Disorder (SAD). We seek to test whether changes in CR and AR underlie the therapeutic effects of CBT and MBSR, which have been shown in the clinical science literature to be effective treatments for SAD. We will examine CR and AR in healthy controls (HCs) and in participants with generalized SAD at baseline, as well as in participants with SAD after they have completed a randomized controlled trial (RCT) with three treatment arms: CBT, MBSR, or Waitlist (WL). This work will address 3 aims: Aim 1 will examine the efficacy of CR and AR in individuals with SAD versus HCs; Aim 2 will investigate the immediate and longer-term impact of CBT versus MBSR for SAD; and Aim 3 will examine treatment-related changes in CR and AR and test whether these changes mediate the effects of CBT versus MBSR. The broad, long-term objective of this research is to contribute to advances in clinical interventions targeting individuals suffering from SAD, as well as a wide range of other anxiety and mood disorders.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosable social anxiety disorder (generalized subtype per DSM-IV-TR criteria)
* aged 21-55
* working fluency in English
* residence in the Bay Area.
* eligible for fMRI scans (right-handed, no metal in body, etc.)

Exclusion Criteria:

* left-handed
* Medication use in the last 3 months
* Pervasive developmental disability
* acute suicide potential
* inability to travel to the treatment site
* schizophrenia or other psychotic disorder
* history of bipolar disorder
* current primary Major Depression
* current substance dependence
* Comorbid diagnoses of Major Depressive or other mood or anxiety disorders are acceptable ONLY if clearly secondary to the diagnosis of social anxiety disorder.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2011-03; Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
Changes in Liebowitz Social Anxiety Scale (LSAS) | from baseline to 1- year following treatment
  The Liebowitz Social Anxiety Scale (LSAS) is a self-report questionnaire which assesses the severity of social anxiety symptoms (Fresco et al., 2001; Liebowitz, 1987). Respondents are asked to rate their level of fear and avoidance to 11 social interaction situations and 13 performance situations. A 4-point Likert-type scale is used for ratings of fear and of avoidance, with a range from 0 (none and never, respectively) to 3 (severe and usually, respectively) for each situation during the past week. Ratings are summed for a total LSAS-SR score (range 0 to 144). The LSAS-SR has demonstrated good reliability and construct validity (Rytwinski et al., 2009).

CONTACTS AND LOCATIONS:
Overall Officials: James J Gross, PhD, Principal Investigator — Stanford University; Philippe R. Goldin, PhD, Study Director — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liebowitz MR. Social phobia. Mod Probl Pharmacopsychiatry. 1987;22:141-73. doi: 10.1159/000414022. No abstract available. PMID 2885745
- [Background] Heimberg RG, Becker RE. Cognitive-behavioral group therapy for social phobia: Basic mechanisms and clinical strategies. Guilford Press; 2002.
- [Background] Hope DA, Heimberg RG, Turk CL. Managing social anxiety: A cognitive-behavioral therapy approach. Treatments That Work; 2010.
- [Background] Kabat-Zinn J. Mindfulness meditation: Health benefits of an ancient Buddhist practice. In D. Goleman & J. Gurin (Eds.), Mind/Body Medicine (pp. 259-275). Yonkers, NY: Consumer Reports Books, 1993.
- [Background] Stahl B, Goldstein E. A mindfulness-based stress reduction workbook. New Harbinger Publications; 2010 Mar 1.
- [Background] American Psychiatric Association. Diagnostic and statistical manual, 4th edn, Text Revision (DSM-IV-TR). American Psychiatric Association, Washington. 2000.
- [Result] Goldin PR, Morrison A, Jazaieri H, Brozovich F, Heimberg R, Gross JJ. Group CBT versus MBSR for social anxiety disorder: A randomized controlled trial. J Consult Clin Psychol. 2016 May;84(5):427-37. doi: 10.1037/ccp0000092. Epub 2016 Mar 7. PMID 26950097
- [Result] Goldin PR, Morrison AS, Jazaieri H, Heimberg RG, Gross JJ. Trajectories of social anxiety, cognitive reappraisal, and mindfulness during an RCT of CBGT versus MBSR for social anxiety disorder. Behav Res Ther. 2017 Oct;97:1-13. doi: 10.1016/j.brat.2017.06.001. Epub 2017 Jun 3. PMID 28654771
- [Derived] Morrison AS, Ustun B, Horenstein A, Kaplan SC, de Oliveira IR, Batmaz S, Gross JJ, Sadikova E, Hemanny C, Pires PP, Goldin PR, Kessler RC, Heimberg RG. Optimized short-forms of the Cognitive Distortions Questionnaire. J Anxiety Disord. 2022 Dec;92:102624. doi: 10.1016/j.janxdis.2022.102624. Epub 2022 Aug 20. PMID 36087565
- [Derived] Goldin PR, Thurston M, Allende S, Moodie C, Dixon ML, Heimberg RG, Gross JJ. Evaluation of Cognitive Behavioral Therapy vs Mindfulness Meditation in Brain Changes During Reappraisal and Acceptance Among Patients With Social Anxiety Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Oct 1;78(10):1134-1142. doi: 10.1001/jamapsychiatry.2021.1862. PMID 34287622
- [Derived] Kuo JR, Zeifman RJ, Morrison AS, Heimberg RG, Goldin PR, Gross JJ. The moderating effects of anger suppression and anger expression on cognitive behavioral group therapy and mindfulness-based stress reduction among individuals with social anxiety disorder. J Affect Disord. 2021 Apr 15;285:127-135. doi: 10.1016/j.jad.2021.02.022. Epub 2021 Feb 8. PMID 33647580
- [Derived] O'Day EB, Butler RM, Morrison AS, Goldin PR, Gross JJ, Heimberg RG. Reductions in social anxiety during treatment predict lower levels of loneliness during follow-up among individuals with social anxiety disorder. J Anxiety Disord. 2021 Mar;78:102362. doi: 10.1016/j.janxdis.2021.102362. Epub 2021 Jan 17. PMID 33486385
- [Derived] Butler RM, O'Day EB, Kaplan SC, Swee MB, Horenstein A, Morrison AS, Goldin PR, Gross JJ, Heimberg RG. Do sudden gains predict treatment outcome in social anxiety disorder? Findings from two randomized controlled trials. Behav Res Ther. 2019 Oct;121:103453. doi: 10.1016/j.brat.2019.103453. Epub 2019 Aug 9. PMID 31430688
- [Derived] Horenstein A, Morrison AS, Goldin P, Ten Brink M, Gross JJ, Heimberg RG. Sleep quality and treatment of social anxiety disorder. Anxiety Stress Coping. 2019 Jul;32(4):387-398. doi: 10.1080/10615806.2019.1617854. Epub 2019 May 13. PMID 31082285
- [Derived] Goldin PR, Moodie CA, Gross JJ. Acceptance versus reappraisal: Behavioral, autonomic, and neural effects. Cogn Affect Behav Neurosci. 2019 Aug;19(4):927-944. doi: 10.3758/s13415-019-00690-7. PMID 30656602
- [Derived] Butler RM, Boden MT, Olino TM, Morrison AS, Goldin PR, Gross JJ, Heimberg RG. Emotional clarity and attention to emotions in cognitive behavioral group therapy and mindfulness-based stress reduction for social anxiety disorder. J Anxiety Disord. 2018 Apr;55:31-38. doi: 10.1016/j.janxdis.2018.03.003. Epub 2018 Mar 9. PMID 29558650